CLINICAL TRIAL: NCT02315651
Title: Efficacy of Combined Treatment With Co-enzyme Q10 and Methylphenidate in Children With Attention Deficit Hyperactivity Disorder
Brief Title: Efficacy of Combined Treatment With CoQ10 and Methylphenidate in Children With Attention Deficit Hyperactivity Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 7636
Record Dates: First submitted 2014-11-03; First posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coenzyme Q10 (Experimental): 30 children aged 6-12 will consume daily a snack containing 60 mg of CoQ10 for 8 weeks.
  Interventions: Dietary Supplement: Coenzyme Q10
- Placebo (Placebo Comparator): 30 children aged 6-12 years will consume an identical snack without CoQ10 for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — A snack containing 60 mg of Coenzyme Q10. The snack contains also dried fruits and nuts, and their content are identical to this of placebo.
  Arms: Coenzyme Q10
Dietary Supplement: Placebo — A snack identical to the trial snack, but without Coenzyme Q10. The snack contains also dried fruits and nuts.
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effects of nutritional supplement co-enzyme Q10 (CoQ10) on methylphenidate-treated ADHD children in a randomized, double-blinded, placebo-controlled prospective study. All eligible patients will undergo randomization and divided into 2 groups: a CoQ10-enriched snack and a placebo snack group. According to power calculation, total of 60 subjects are expected to participate in the study. After the screening of eligibility (up to 14 days), the study is divided into three phases: pre-treatment (first assessment) phase (up to 14 days), treatment phase 8 weeks of treatment, and post-treatment phase. Screening: each participant will undergo screening for protocol eligibility within 14 days (two weeks) of recruitment. Subjects who meet all the inclusion criteria and signed an approved informed consent (both parents and the child) will be enrolled.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effects of nutritional supplement co-enzyme Q10 (CoQ10) on methylphenidate-treated ADHD children in a randomized, double-blinded, placebo-controlled prospective study. All eligible patients will undergo randomization and divided into 2 groups: a CoQ10-enriched snack and a placebo snack group. According to power calculation, total of 60 subjects are expected to participate in the study. After the screening of eligibility (up to 14 days), the study is divided into three phases: pre-treatment (first assessment) phase (up to 14 days), treatment phase 8 weeks of treatment, and post-treatment phase. Screening: each participant will undergo screening for protocol eligibility within 14 days (two weeks) of recruitment. Subjects who meet all the inclusion criteria and signed an approved informed consent (both parents and the child) will be enrolled.

Pre-treatment period (1-st phase): for the purpose of the first assessment, participants' parents will receive Conner's questionnaire for filling by parents and teachers. The first nutritional assessment will be undertaken using 24-h recall assessment.

Treatment period (2-st phase): randomization and treatment. After randomization to 2 groups, CoQ10 and placebo groups, the participants' parents will receive either CoQ10-enriched or placebo snack for 8 weeks (2 months) period. The participants and their parents will be instructed to consume the snack daily. During the study the subjects will manage with their methylphenidate treatment as indicated by their neurologist.

Post-treatment assessment (3-rd phase): At the end of the study period, an additional assessment identical to this of the pre-treatment will be taken to evaluate subjects' response to the snacks.

Statistical analysis (4-th phase): At the end of the study, statistical analysis will be undertaken. Statistical difference between two groups in their pre-treatment and post-treatment behavioral and nutritional response will serve as an evidence for the efficacy of the supplement being used. All data will be documented in patient charts and individual computerized case report form .

The duration of the study is expected to be 2 years.

ELIGIBILITY:
Inclusion Criteria:

Children aged 6-12. Diagnosed as ADHD according to DSM4 At least 3 months treated with methylphenidate Informed consent of a parent and agreement of a teacher for participation in the trial -

Exclusion Criteria:

Adolescent girls after more than 3 menses History or current diagnosis of systemic diseases, diabetes, thyroid abnormalities or problems with neural system, such as epilepsy or brain tumor.

Children with other psychiatric disorders, as diagnosed according to DSM4. Children with a risk to suicide. Using of psychiatric medications other then methylphenidate. Using of dietary supplements at least 4 weeks before enrollment. History of abuse of alcohol or drugs according to DSM4. Consuming of above 250 mg of caffeine. Allergy for one of the snack's ingredients. Use of drugs for chronic diseases

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of an effect of coenzyme CoQ10 on behavioral aspects of methylphenidate- treated ADHD children | 60 days
  The evaluation will be executed with Conners score

SECONDARY OUTCOMES:
Evaluation of an effect of coenzyme Q10 on nutritional behavior of methylphenidate- treated ADHD children | 60 days
  The evaluation will be executed with 24-h recall and measuring of BMI

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Straussberg, Prof., Principal Investigator — Schneider children's medical center of Israe
Locations (1):
- Schneider children's medical center of Israel, Petah Tikva, Israel